CLINICAL TRIAL: NCT07221175
Title: Evaluation of Radiation Dose of the Operator Using an Ultra-Low Dose 3.75 Fluoroscopic Pulse Rate Versus Standard 7.5 Fluoroscopic Pulse Rate Performing Coronary Angiography Via Right Radial Artery Approach: A Randomized Clinical Trial.
Brief Title: Operator Radiation Dose Using Ultra-Low Fluoroscopic Pulse Rate Versus Standard In Performing Coronary Angiography Via Right Radial Artery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maimonides Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2024-12-08-MMC
Record Dates: First submitted 2025-10-20; First posted 2025-10-27 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Radiation Exposure; Radiation Exposure to Operator
Keywords: Radiation exposure; Radial approach; Cardiac catheterization; Coronary angiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Ultra-low dose 3.75 fluoroscopic pulses per second (Experimental): Radiation exposure to the operator performing diagnostic coronary angiography via right radial artery approach utilizing an ultra-low dose fluoroscopic pulse rate of 3.75 frames per second
  Interventions: Radiation: Ultra low dose fluoroscopic pulse rate
- Standard low-dose 7.5 fluoroscopic pulses per second (Active Comparator): Radiation exposure to the operator performing diagnostic coronary angiography via right radial artery approach utilizing a standard low dose fluoroscopic pulse rate of 7.5 frames per second
  Interventions: Radiation: Standard low dose fluoroscopic pulse rate

INTERVENTIONS:
Radiation: Ultra low dose fluoroscopic pulse rate — Ultra low dose 3.75 fluoroscopic pulses per second
  Arms: Ultra-low dose 3.75 fluoroscopic pulses per second
Radiation: Standard low dose fluoroscopic pulse rate — Standard low dose 7.5 fluoroscopic pulses per second
  Arms: Standard low-dose 7.5 fluoroscopic pulses per second

SUMMARY:
The goal of this randomized clinical trial is to determine if there can be reduction in the radiation exposure to the cardiologist performing a coronary angiogram via a right radial artery approach by using a lower fluoroscopic pulse rate. Researchers will compare the radiation dose received by the primary operator using an ultra-low fluoroscopic pulse rate of 3.75 frames per second compared to the standard low pulse rate of 7.5 frames per second. Participating operators will wear multiple dosimeters, and the difference of radiation exposure will be measured.

DETAILED DESCRIPTION:
Radiation exposure is one of the most adverse occupational hazards faced by interventional cardiologists. Though there have been many technologic advances over the years which have reduced the amount of radiation received by the operating physician, there is still a non-negligible amount of radiation that the operator is exposed to. The reduction of fluoroscopic pulse rate during cardiac catheterization has been shown to reduce both operator and patient radiation exposure. Current standard of practice is still to use up to 15 frames per second of fluoroscopy during coronary angiogram, with some centers adapting a low-dose 7.5 frames per second as standard. However, an ultra-low dose of 3.75 frames per second is not often utilized.

The right radial artery is the preferred access route for interventional cardiologists; they are familiar with working from the right side of the catheterization table and this is how standard laboratory equipment has historically been configured. This trial will determine if using an ultra-low fluoroscopic pulse rate of 3.75 frames per second will reduce both physician and patient radiation exposure, compared to the low-dose pulse rate of 7.5 frames per second being utilized in coronary angiography performed via right radial approach.

Procedures will be randomized to be performed with either the 3.75 frames per second or 7.5 frames per second. Only diagnostic procedures performed via right radial approach will be included. The primary operators will be equipped with radiation dosimeters at the level of the thorax and the right and left eyes. Both cumulative and normalized levels of radiation will be assessed per individual procedure performed via right radial approach. As a secondary outcome, the difference in the radiation exposure (dose-area product and milligray) of the patient will also be measured.

ELIGIBILITY:
Inclusion Criteria:

* Operators using the right radial approach as a primary access site
* Patients of any sex and gender.
* Patients Age > 18 years old.
* Patients undergoing diagnostic coronary angiogram from in-patient and out-patient settings from the right radial artery approach

Exclusion Criteria:

* All operators performing cardiac catheterization from an access point other than the right radial artery
* All patients undergoing cardiac catheterization from an access point other than the right radial artery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 338 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Radiation exposure to the operator | Periprocedural per each individual procedure
  To observe the difference of radiation exposure (cumulative and normalized) at the level of the thorax, left eye, and right eye of the operator comparing a 7.5 fluoroscopic pulse rate and an ultra-low 3.75 fluoroscopic pulse rate

SECONDARY OUTCOMES:
Radiation exposure to patient | Periprocedural per each individual procedure
  To observe the difference of radiation exposure to the patient (dose area product, milligray) comparing a 7.5 fluoroscopic pulse rate and an ultra-low 3.75 fluoroscopic pulse rate

CONTACTS AND LOCATIONS:
Overall Officials: Bilal A Malik, MD, Principal Investigator — Maimonides Medical Center
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Radiation exposure measured per dosimeter per procedure for the operators, and patient radiation exposure per procedure.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be available following termination of the data collection and analysis (date to be determined, estimate 2/1/2027) for up to 3 years (2/1/2030).
Access Criteria: IPD can be requested by e-mailing the primary contact point.

REFERENCES:
- [Result] Agarwal S, Parashar A, Ellis SG, Heupler FA Jr, Lau E, Tuzcu EM, Kapadia SR. Measures to reduce radiation in a modern cardiac catheterization laboratory. Circ Cardiovasc Interv. 2014 Aug;7(4):447-55. doi: 10.1161/CIRCINTERVENTIONS.114.001499. Epub 2014 Aug 5. PMID 25097198
- [Result] Abdelaal E, Plourde G, MacHaalany J, Arsenault J, Rimac G, Dery JP, Barbeau G, Larose E, De Larochelliere R, Nguyen CM, Allende R, Ribeiro H, Costerousse O, Mongrain R, Bertrand OF; Interventional Cardiologists at Quebec Heart-Lung Institute. Effectiveness of low rate fluoroscopy at reducing operator and patient radiation dose during transradial coronary angiography and interventions. JACC Cardiovasc Interv. 2014 May;7(5):567-74. doi: 10.1016/j.jcin.2014.02.005. Epub 2014 Apr 16. PMID 24746649